CLINICAL TRIAL: NCT06522412
Title: The Effects of Jing-Si Herbal Tea Liquid Packets and Jing-Si Herbal Tang Heng Power Drink on Metabolism and Inflammation in Patients With Cardiovascular Diseases
Brief Title: The Effects of Jing-Si Herbal Tea Liquid Packets and Jing-Si Herbal Tang Heng Power Drink
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Chang Huai Ren, Principal Investigator, Buddhist Tzu Chi General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB 113-012-A
Record Dates: First submitted 2024-06-20; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Inflammatory Marker; Gut Microbiome; Trimethylamine N-oxide; HbA1c; Atherosclerosis
Keywords: trimethylamine N-oxide; gut microbiome; cardiovascular disease; atherosclerosis
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TL_TH (Experimental): The participants takeJING SI HERBAL TEA LIQUID PACKETS first for 12 weeks and then wash-out for 12 weeks, and then take JING SI HERBAL TANG HENG POWDER DRINK for 12 weeks.
  Interventions: Dietary Supplement: JING SI HERBAL TEA LIQUID PACKETS; Dietary Supplement: JING SI HERBAL TANG HENG POWDER DRINK
- TH_TL (Active Comparator): The participants take JING SI HERBAL TANG HENG POWDER DRINK first for 12 weeks and then wash-out for 12 weeks, and then take JING SI HERBAL TEA LIQUID PACKETS for 12 weeks.
  Interventions: Dietary Supplement: JING SI HERBAL TEA LIQUID PACKETS; Dietary Supplement: JING SI HERBAL TANG HENG POWDER DRINK

INTERVENTIONS:
Dietary Supplement: JING SI HERBAL TEA LIQUID PACKETS — JING SI HERBAL TEA LIQUID PACKETS contains: eight herbal ingredients, primarily including dwarf lilyturf, houttuynia, balloon flower, siegesbeckia, licorice, mugwort, perilla leaf, and chrysanthemum. These eight Taiwanese native herbs are known for their abilities to moisturize, disperse cold, relieve lung congestion, dissolve phlegm, remove dampness, and clear heat.
Dietary Supplement: JING SI HERBAL TANG HENG POWDER DRINK — JING SI HERBAL TANG HENG POWDER DRINK contains: Based on the eight herbal ingredients of Jingsi Herbal Drink Concentrate, this drink additionally includes pumpkin powder and bitter melon extract powder. (Ingredients: siegesbeckia, Jingsi complex herbal powder (dextrin fiber, herbal extracts (mugwort, siegesbeckia, dwarf lilyturf, houttuynia, balloon flower, licorice, perilla leaf, chrysanthemum)), pumpkin powder, bitter melon extract powder (bitter melon extract (containing bitter melon peptides), maltodextrin), black pepper, chromium nicotinate complex (chromium nicotinate, sodium chloride)).

SUMMARY:
Through empirical research evaluating the effects of "JING SI HERBAL TEA LIQUID PACKETS" and "JING SI HERBAL TANG HENG POWDER DRINK" as adjunctive treatments for various cardiovascular diseases, we aim to provide sufficient evidence to address the following questions:

1. Can "JING SI HERBAL TEA LIQUID PACKETS" and "JING SI HERBAL TANG HENG POWDER DRINK" significantly improve various inflammatory responses involved in the process of atherosclerosis, thereby enhancing the prognosis of patients with acute coronary syndrome and chronic ischemic heart disease?
2. Can "JING SI HERBAL TEA LIQUID PACKETS" and "JING SI HERBAL TANG HENG POWDER DRINK" provide a healthy and effective adjunctive therapy for patients with hypertension, diabetes, and hyperlipidemia by lowering blood pressure (potentially related to known ACE2 receptors), blood glucose levels (including the improvement of pancreatic β-cell insulin secretion capacity and cellular insulin utilization efficiency), and cholesterol levels?
3. Can "JING SI HERBAL TEA LIQUID PACKETS" and "JING SI HERBAL TANG HENG POWDER DRINK" influence the prognosis of various diseases, including the most critical cardiovascular conditions such as acute coronary syndrome and chronic ischemic heart disease, by altering the human gut microbiota?
4. Can "JING SI HERBAL TEA LIQUID PACKETS" and "JING SI HERBAL TANG HENG POWDER DRINK" improve renal indicators such as BUN, creatinine, UACR, and eGFR, thereby protecting the kidneys and reducing complications like microalbuminuria?

DETAILED DESCRIPTION:
The Jing-Si Herbal Drink is composed of eight native Taiwanese herbal ingredients: mugwort, fishwort, houttuynia, dwarf lilyturf, balloon flower, perilla leaf, chrysanthemum, and licorice. These ingredients are known for their properties to clear heat, dispel cold, ventilate the lungs, transform phlegm, and eliminate dampness. Preliminary cell and animal studies have demonstrated that this drink can block the binding of the novel coronavirus (SARS-CoV-2) to cells and reduce cellular penetration, thereby preventing the virus from entering the cells. Recently, the Jing-Si Herbal Drink in powder form, known as "Jing-Si Herbal Drink Concentrate Powder," received an export-specific license from the Ministry of Health and Welfare. A research team from Taipei Tzu Chi Hospital has confirmed that combining standard treatment with Jing-Si Herbal Drink provides good clinical protective effects and safety for patients with mild to moderate COVID-19.

Angiotensin-converting enzyme 2 (ACE2), encoded by the ACE2 gene located on the X chromosome, regulates blood pressure and endocrine functions by clearing the vasopressor angiotensin II (Ang II), thereby allowing blood vessels to relax. Studies have shown that the human ACE2 receptor is the gateway for the novel coronavirus (SARS-CoV-2) to enter cells. Both the novel coronavirus and the SARS coronavirus must bind to the ACE2 receptor via their spike proteins to enter cells and replicate extensively, leading to pathogenicity. It is therefore reasonable to hypothesize that the Jing-Si Herbal Drink may block the binding of the novel coronavirus (SARS-CoV-2) to cells by regulating the ACE2 receptor.

Recently, the basic medical research team on herbal drinks at Hualien Tzu Chi Hospital has demonstrated through animal experiments that the Jing-Si Herbal Drink has significant anti-aging protective effects on cardiovascular and metabolic functions in aged rats (24-month-old WKY rats). Additionally, a preliminary analysis conducted by Professor Hong-Chih Han's laboratory at the Hualien Tzu Chi Hospital's Innovation and Research Center revealed that various aspects of immune function were positively affected by the Jing-Si Herbal Drink. It was observed that IFN-γ levels in the blood of subjects significantly increased 48-96 hours after consumption of the Jing-Si Herbal Drink, suggesting that it plays an important role in immune regulation.

The Jing-Si Abode Herbal Research and Development Team has built upon the original Jing-Si Herbal Drink formula to create a new generation of herbal beverage: Jing-Si Herbal Sugar-Balance Beverage. This new formula incorporates pumpkin powder and bitter melon extract powder (containing bitter melon peptides) in addition to the eight original herbal ingredients of the concentrated herbal drink. It is expected to provide enhanced protection for blood sugar and lipid metabolism as well as immune function. Recently, the basic medical research team on herbal drinks at Hualien Tzu Chi Hospital conducted animal experiments that preliminarily confirmed the superior blood sugar-lowering effects of the Jing-Si Herbal Sugar-Balance Beverage formula in diabetic rats compared to the original Jing-Si Herbal Drink formula and the drug Metformin.

The investigators will leverage the professional care provided by clinical physicians and the analytical research capabilities of our basic laboratory to collaboratively evaluate the effects of "Jing-Si Herbal Drink Concentrate" and "Jing-Si Herbal Drink Sugar-Balance Beverage" as adjunctive treatments for patients with various cardiovascular diseases. The investigators aim to not only improve the quality of life for these patients but also achieve beneficial outcomes in treating some clinically challenging diseases and symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-75 years.
2. Diagnosed with any of the following diseases:

(1) Hypertension (2) Hyperlipidemia (3) Diabetes (4) Ischemic heart disease"

Exclusion Criteria:

1. History of cancer.
2. Subjects with severe or poorly controlled chronic diseases as determined by the principal investigator.
3. Poor renal function (eGFR <40 ml/min/1.73m²).
4. Pregnant or breastfeeding at the time of screening.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Effect of intervention on lipid profile | Baseline, 4 and 12 weeks after intervention is given.
  TCH、TG、HDL-C、LDL-C
Effect of blood uric acid on Cardiovascular Disease and body inflammation status | Baseline, 4 and 12 weeks after intervention is given.
  Uric acid
Effect of intervention on fasting sugar | Baseline, 4 and 12 weeks after intervention is given.
  Glu-AC
To evaluate the metabolic health | Baseline, 4 and 12 weeks after intervention is given.
  Uric acid
Long term blood sugar status | Baseline, 4 and 12 weeks after intervention is given.
  HbA1C
Homeostatic model assessment (HOMA) of insulin resistance | Baseline, 4 and 12 weeks after intervention is given.
  HOMA-IR is calculated by insulin level and Glu-AC
Inflammation biomarkers | Baseline, 4 and 12 weeks after each intervention is given.
  hs-C-reactive protein
The hematological parameter for systemic inflammation and stress | Baseline, 4 and 12 weeks after each intervention is given.
  neutrophil-to-lymphocyte ratio, platelet-to-lymphocyte ratio
proinflammtory marker | Baseline, 4 and 12 weeks after each intervention is given.
  Glyc-A
Liver function | Baseline, 4 and 12 weeks after each intervention is given
  GOT、GPT
Kidney function | Baseline, 4 and 12 weeks after each intervention is given
  BUN、Cre、eGFR(Calculated by age and Cre)
Evaluation of activity of gut microbiome | Baseline, 4 and 12 weeks after each intervention is given
  TMA、TMAO
The concentration of the product of gut microbiome | Baseline, 4 and 12 weeks after each intervention is given
  SCFA (short-chain fatty acid)
Analysis of Gut Microbiota in Stool Samples Using 16S rRNA Sequencing | Stool samples will be collected at baseline (prior to intervention) and at 12 months post-intervention to assess changes in gut microbiota composition and abundance.
  This study aims to analyze the gut microbiota in stool samples to assess changes in microbial composition and abundance following the intervention. The primary objective is to determine if the intervention lead to significant shifts in the diversity and relative proportions of gut bacteria
Body fat composition | Baseline, 4 and 12 weeks after each intervention is given
  BMI(calculated y weight and height)
To evaluate the distribution of body fat | Baseline, 4 and 12 weeks after each intervention is given
  Waist-to-Hip Ratio
Effect of intervention on blood pressure control | Baseline, 4 and 12 weeks after each intervention is given
  blood pressure
Measurement of overall immune function and response to infection or inflammation | Baseline, 4 and 12 weeks after each intervention is given
  WBC
Evaluate the immune system function | Baseline, 4 and 12 weeks after each intervention is given
  CD3、CD4、CD8、CD56
Assessment of leukocyte activation | Baseline, 4 and 12 weeks after each intervention is given
  CD11b
To evaluates the body's ability to fight tumors and infections. | Baseline, 4 and 12 weeks after each intervention is given
  NK cells
To assess immune activation and the ability to present antigens to T cells | Baseline, 4 and 12 weeks after each intervention is given
  HLA-DR
Assessment of immune response | Baseline, 4 and 12 weeks after each intervention is given
  IFN-gamma、IL-6
Marker of inflammation | Baseline, 4 and 12 weeks after each intervention is given
  TNF-alpha

CONTACTS AND LOCATIONS:
Locations (1):
- Hualien Tzu Chi Hospital, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: No